CLINICAL TRIAL: NCT00044083
Title: Randomized, Double-Blinded, Placebo Controlled Study of the Effects of Tolcapone and Entacapone on Cognitive Function in Patients With Schizophrenia and Normal Controls Based on COMT Genotype
Brief Title: Clinical Trial of Tolcapone for Cognition in Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Scientific Director request to use resources for other studies
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 020239; 02-M-0239 (Other: Clinicaltrials.gov); NCT00044083 (Other: Clinicaltrials.gov)
Record Dates: First submitted 2002-08-16; First posted 2002-08-19 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
Keywords: Catecholamines; Dopamine; Clinical Trial; fMRI; PFC; Vitamin B2; Riboflavin; Tolcapone; Placebo; Normal Volunteers; Schizophrenia; Healthy Volunteers; HV
MeSH Terms: conditions — Schizophrenia | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Placebo one week
  Interventions: Other: Placebo
- Tolcapone Arm (Active Comparator): Tolcapone one week
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Other: Placebo — Placebo: One capsule 3 times a day from Day 1 to Day 7
  Arms: Placebo Arm
Drug: Tolcapone — Tolcapone: One capsule 3 times a day from Day 1 to Day 7
  Other Names: Tasmar
  Arms: Tolcapone Arm

SUMMARY:
This study will evaluate whether Tolcapone improves cognition in healthy volunteers as well as patients with schizophrenia. Talcapone is a drug that has been FDA approved for Attention Deficit Disorder and allegedly increase the amount of the neurotransmitter dopamine in the frontal cortex of the brain.

...

DETAILED DESCRIPTION:
Psychopharmacological modulation of the catecholaminergic system can enhance some aspects of cognitive function. For example, COMT inhibitors can slightly improve working memory/executive function. Differences in the response between individuals might be related to a number of factors, including variations in the genes. The recent finding that a polymorphism in the catechol-o-methyl-transferase (COMT) gene, which produces a 4 fold change in enzyme activity, accounts for 4 percent of the variance in performance of working memory tasks in humans suggest that COMT genotype may predict response to COMT inhibitors. In the present investigation our goal is to examine, in normal controls and patients with schizophrenia, the effect of a centrally acting (tolcapone) and of a peripherally acting (entacapone) COMT inhibitor on cognitive function. We predict that both normal controls and patients with schizophrenia with the val/val genotype will have a significant, though transient, improvement in working memory in subjects treated with tolcapone but not in those treated with entacapone. Furthermore, in conjunction with other NIMH imaging protocols, we would like to examine the neurophysiological correlates related to working memory. We predict, in tolcapone treated subjects, improved measures in prefrontal 'efficiency' in subjects and patients specifically with the val/val genotype. The present protocol will provide new insights on the importance of this genetic polymorphism in the regulation of aminergic-controlled cognitive function in normal individuals. Furthermore, this protocol will test whether COMT inhibitors offer a new treatment-based on genotype - for cognitive impairment in schizophrenia. No IND is required for the present study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Prior participation under NIH protocol number 95-M-0150, or new normal volunteers or schizophrenic patients that meet criteria for NIH protocol number 95-M-0150 (NCT00001486).
  2. No Axis I or Axis II diagnosis in normal volunteers.
  3. Age range: 18-50 years.

EXCLUSION CRITERIA:

1. Normal volunteers with an Axis I or Axis II disorder obtained either from prior SCID interview in Protocol 95-M-0150 or through a screening interview will be excluded.
2. Subjects with a history of cardiovascular disease, liver disease and other medical illnesses, and untreated or uncontrolled hypertension will be excluded. An electrocardiogram, blood pressure, pulse rate and metabolic panel including LFTs will be checked on all subjects prior to participation in the study. Individuals with persistent tardive dyskinesia or abnormal LFTs, or individuals with significant history of alcoholism or liver enzyme elevation will be excluded from the study.
3. Schizophrenic patients taking clozapine, a COMT inhibitor, any illicit drugs of abuse, or MAO inhibitors will be excluded.
4. Normal control subjects taking any medications other than occasional NSAI will be excluded.
5. Pregnant women. Women of childbearing potential will undergo a urine pregnancy test the day the study initiates and screened by history for the possibility of pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2002-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Apud, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Aksoy S, Klener J, Weinshilboum RM. Catechol O-methyltransferase pharmacogenetics: photoaffinity labelling and western blot analysis of human liver samples. Pharmacogenetics. 1993 Apr;3(2):116-22. doi: 10.1097/00008571-199304000-00008. PMID 8518836
- [Background] Andreasen NC, Arndt S, Cizadlo T, O'Leary DS, Watkins GL, Ponto LL, Hichwa RD. Sample size and statistical power in [15O]H2O studies of human cognition. J Cereb Blood Flow Metab. 1996 Sep;16(5):804-16. doi: 10.1097/00004647-199609000-00005. PMID 8784225
- [Background] Arnsten AF. Catecholamine regulation of the prefrontal cortex. J Psychopharmacol. 1997;11(2):151-62. doi: 10.1177/026988119701100208. PMID 9208378
- [Derived] Magalona SC, Rasetti R, Chen J, Chen Q, Gold I, Decot H, Callicott JH, Berman KF, Apud JA, Weinberger DR, Mattay VS. Effect of tolcapone on brain activity during a variable attentional control task: a double-blind, placebo-controlled, counter-balanced trial in healthy volunteers. CNS Drugs. 2013 Aug;27(8):663-73. doi: 10.1007/s40263-013-0082-x. PMID 23794107
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-M-0239.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with schizophrenia were recruited through families, physicians and community organizations. Healthy volunteers were recruited through the NIH Normal Volunteers Office. Subjects first participated in Protocol # 95-M-0150 to obtain genotype data. If eligible after the study, they were invited to participate in the Tolcapone protocol.
Groups:
- Placebo First Then Tolcapone: Placebo one week first:
  Tolcapone 200 mg second:
- Tolcapone First, Then Placebo: Tolcapone one week:
  Placebo one week second:
Period: First Intervention (One Week)- HV's
Arm/Group | Placebo First Then Tolcapone | Tolcapone First, Then Placebo
Started | 74 | 73
Completed | 64 | 66
Not Completed | 10 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Not follow directions | 2 | 2
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Used illegal drugs | 1 | 0
Not completed — Abnormal MRI | 0 | 1
Not completed — Drank while on protocol | 0 | 1
Period: Second Intervention (One Week) HV's
Arm/Group | Placebo First Then Tolcapone | Tolcapone First, Then Placebo
Started | 64 | 66
Completed | 64 | 66
Not Completed | 0 | 0
Period: First Intervention (One Week) Patients
Arm/Group | Placebo First Then Tolcapone | Tolcapone First, Then Placebo
Started | 31 | 32
Completed | 30 | 30
Not Completed | 1 | 2
Not completed — Not follow directions | 0 | 2
Not completed — Used illegal drug | 1 | 0
Period: Second Intervention (One Week) Patients
Arm/Group | Placebo First Then Tolcapone | Tolcapone First, Then Placebo
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: These numbers represent the total number of subjects (HV's+patients) plus HV's and patients separately that completed the first and second arm of the protocol.
Groups:
- Healthy Volunteers; Patients: Tolcapone 200 mg 1 week:Wash Out 1 week:Placebo 1 week: (or vice versa)
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Patients | Total
Number analyzed (Participants) | 130 | 59 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 130 | 59 | 189
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.1) | 26.9 (6.8) | 32.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 18 | 77
  Male | 71 | 41 | 112
Region of Enrollment [Number; unit: participants]
  United States | 130 | 59 | 189

OUTCOME MEASURES:

1. Primary Outcome: N-Back Task Performance
Description: Working Memory was measured in HVs and patients with schizophrenia after a 7-day treatment with Tolcapone or placebo in a double-blind, cross-over fashion. The working memory was quantified by taking the number of trials entered correctly divided by the total number of trials multiplied by 100. Values range from 0 to 100. Zero indicates the poorest performance while 100 indicates perfect performance.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 147 HV's recruited, 8 left after signing consents, 8 excluded for other reasons, 57 excluded for excessive motion, inferior quality or not completion. 63 patients recruited, 4 removed for different reasons, 26 excluded from image analyses for not completing the second phase of the study, excessive motion or bad image quality.
Measure: Mean (Standard Error); unit: % of Correct Trials
Groups:
- Healthy Volunteer on Placebo: Placebo Days 1-7, Healthy voluntee
- Healthy Volunteer Tolcapone; Patients on Tolcapone: Day 1: Tolcapone 100 mg tid, Days 2-7: Tolcapone 200 mg tid
- Patient on Placebo: Placebo Days 1-7, Patient
Arm/Group | Healthy Volunteer on Placebo | Healthy Volunteer Tolcapone | Patient on Placebo | Patients on Tolcapone
Number analyzed (Participants) | 74 | 74 | 33 | 33
% of Correct Trials | 86.10 (1.13) | 85.50 (1.10) | 76.21 (2.31) | 80.94 (1.90)
Statistical Analysis 1: Comparison: Healthy Volunteer on Placebo vs Patient on Placebo; Test type: Other; p < 0.0001, ANOVA — Diagnosis effect on placebo
Statistical Analysis 2: Comparison: Patient on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.0034, ANOVA — Drug Effect on Patients

2. Primary Outcome: N-Back Task Activation Diagnosis Effect
Description: Activation beta values (N-Back vs. 0-Back) were extracted within the Main Effect of Diagnosis cluster around the peak (p < 0.05 uncorrected) from the contrast maps in the Placebo condition. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 74 Healthy Volunteers and 33 Patients with Schizophrenia
Measure: Mean (Standard Error); unit: beta value
Groups:
- Healthy Volunteer on Placebo: Placebo Days 1-7, Healthy Voluntreers
- Patient on Placebo: Placebo Days 1-7, Patients
Arm/Group | Healthy Volunteer on Placebo | Patient on Placebo
Number analyzed (Participants) | 74 | 33
beta value
  Right DLPFC | 0.15 (0.02) | 0.20 (0.03)
  Left DLPFC | 0.18 (0.02) | 0.23 (0.03)
Statistical Analysis 1: Comparison: Healthy Volunteer on Placebo vs Patient on Placebo; Test type: Other; p < 0.0001, ANOVA — Diagnosis Effect on Placebo in right DLPFC
Statistical Analysis 2: Comparison: Healthy Volunteer on Placebo vs Patient on Placebo; Test type: Other; p = 0.014, ANOVA — Diagnosis Effect of Placebo in left DLPFC

3. Primary Outcome: N-Back Task Activation Drug Effect
Description: Activation beta values (N-Back vs. 0-Back) extracted within the Main Effect of Drug cluster around the peak (p < 0.05 uncorrected) from the contrast maps across both groups. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 74 Healthy Volunteers and 33 Patients with Schizophrenia
Measure: Mean (Standard Error); unit: beta value
Groups:
- Healthy Volunteers on Placebo: Placebo Days 1-7, Healthy Volunteers
- Healthy Volunteers on Tolcapone; Patients on Tolcapone: Tolcapone 100 mg TID on Day 1, 200 mg TID Days 2-7.
- Patients on Placebo: Placebo Days 1-7, Patients
Arm/Group | Healthy Volunteers on Placebo | Healthy Volunteers on Tolcapone | Patients on Placebo | Patients on Tolcapone
Number analyzed (Participants) | 74 | 74 | 33 | 33
beta value
  Right DLPFC | 0.09 (0.03) | 0.11 (0.02) | 0.12 (0.04) | 0.07 (0.03)
  Left DLPFC | 0.27 (0.04) | 0.25 (0.04) | 0.23 (0.05) | 0.09 (0.06)
Statistical Analysis 1: Comparison: Healthy Volunteers on Placebo vs Healthy Volunteers on Tolcapone vs Patients on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.05, ANOVA — Drug Effect across both groups in left DLPFC
Statistical Analysis 2: Comparison: Healthy Volunteers on Placebo vs Healthy Volunteers on Tolcapone vs Patients on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.32, ANOVA — Drug Effect across both groups in right DLPFC

4. Primary Outcome: N-Back Task Activation in DLPFC in Patients With Schizophrenia
Description: Activation Beta values (N-Back vs. 0-Back) extracted within the Effect of Drug cluster around the peak (p < 0.05 uncorrected) from the contrast maps in patients with schizophrenia. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 33 Patients with Schizophrenia
Measure: Mean (Standard Error); unit: beta value
Groups:
- Patients on Tolcapone: Day 1 Tolcapone 100 mg tid, days 2-7 Tolcapone 200 mg tid, Patients
Arm/Group | Patients on Placebo | Patients on Tolcapone
Number analyzed (Participants) | 33 | 33
beta value
  Right DLPFC | 0.26 (0.02) | 0.24 (0.018)
  Left DLPFC | 0.25 (0.02) | 0.23 (0.02)
Statistical Analysis 1: Comparison: Patients on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.05, t-test, 1 sided — The Effect of Drug on Patients with Schizophrenia in right DLPFC
Statistical Analysis 2: Comparison: Patients on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.078, t-test, 1 sided — Effect of Drug on Patients with Schizophrenia in left DLPFC

5. Primary Outcome: N-Back Task Activation in Healthy Volunteers
Description: Activation Beta values (N-Back vs. 0-Back) extracted within the Effect of Drug cluster around the peak (p < 0.05 uncorrected) from the contrast maps in Healthy Volunteers. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 74 Healthy Volunteers
Measure: Mean (Standard Error); unit: beta value
Groups:
- Healthy Volunteer on Placebo: Placebo Days 1-7, Healthy Volunteer
- Healthy Volunteer on Tolcapone: Day 1 Tolcapone 100 mg tid, days 2-7 Tolcapone 200 mg tid
Arm/Group | Healthy Volunteer on Placebo | Healthy Volunteer on Tolcapone
Number analyzed (Participants) | 74 | 74
beta value
  Right DLPFC | 0.09 (0.03) | 0.11 (0.02)
  Left DLPFC | 0.38 (0.03) | 0.36 (0.03)
Statistical Analysis 1: Comparison: Healthy Volunteer on Placebo vs Healthy Volunteer on Tolcapone; Test type: Other; p = 0.05, t-test, 1 sided — Drug Effect on Healthy Volunteers in left DLPFC
Statistical Analysis 2: Comparison: Healthy Volunteer on Placebo vs Healthy Volunteer on Tolcapone; Test type: Other; p = 0.73, t-test, 1 sided — Drug Effect on Healthy Volunteers in right DLPFC

6. Primary Outcome: N-Back Task Activation Genotype Effect in Healthy Volunteers
Description: Activation beta values (N-Back vs. 0-Back) extracted within the Effect of Genotype cluster around the peak (p < 0.05 uncorrected) in right and left DLPFC from the contrast maps in Healthy Volunteers. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Measure: Mean (Standard Error); unit: beta value
Groups:
- Healthy Volunteer COMT Val/Val Genotype on Placebo: Placebo Days 1-7, Healthy Volunteer COMT Val/Val Genotype
- Healthy Volunteer COMT Val/Met Genotype on Placebo: Placebo Days 1-7, Healthy Volunteer COMT Val/Met Genotype
- Healthy Volunteers COMT Met/Met Genotype on Placebo: Placebo Days 1-7, Healthy Volunteers COMT Met/Met Genotype
- Healthy Volunteer COMT Val/Val Genotype on Tolcapone: Day 1: Tolcapone 100 mg tid, Days 2-7: Tolcapone 200 mg tid Healthy Volunteer COMT Val/Val Genotype
- Healthy Volunteer COMT Val/Met Genotype on Tolcapone: Day 1: Tolcapone 100 mg tid, Days 2-7: Tolcapone 200 mg tid Healthy Volunteer COMT Val/Met Genotype
- Healthy Volunteer COMT Met/Met Genotype on Tolcapone: Day 1: Tolcapone 100 mg tid, Days 2-7: Tolcapone 200 mg tid Healthy Volunteer COMT Met/Met Genotype
Arm/Group | Healthy Volunteer COMT Val/Val Genotype on Placebo | Healthy Volunteer COMT Val/Met Genotype on Placebo | Healthy Volunteers COMT Met/Met Genotype on Placebo | Healthy Volunteer COMT Val/Val Genotype on Tolcapone | Healthy Volunteer COMT Val/Met Genotype on Tolcapone | Healthy Volunteer COMT Met/Met Genotype on Tolcapone
Number analyzed (Participants) | 24 | 29 | 21 | 24 | 29 | 21
beta value
  Right DLPFC | 0.22 (0.03) | 0.23 (0.03) | 0.14 (0.04) | 0.22 (0.03) | 0.25 (0.03) | 0.15 (0.04)
  Left DLPFC | 0.14 (0.03) | 0.19 (0.03) | 0.10 (0.03) | 0.14 (0.03) | 0.18 (0.03) | 0.09 (0.04)
Statistical Analysis 1: Comparison: Healthy Volunteer COMT Val/Val Genotype on Placebo vs Healthy Volunteer COMT Val/Met Genotype on Placebo vs Healthy Volunteers COMT Met/Met Genotype on Placebo vs Healthy Volunteer COMT Val/Val Genotype on Tolcapone vs Healthy Volunteer COMT Val/Met Genotype on Tolcapone vs Healthy Volunteer COMT Met/Met Genotype on Tolcapone; Test type: Other; p < 0.0001, ANOVA; Main Effect of Genotype across both Placebo and Tolcapone in right DLPFC
Statistical Analysis 2: Comparison: Healthy Volunteer COMT Val/Val Genotype on Placebo vs Healthy Volunteer COMT Val/Met Genotype on Placebo vs Healthy Volunteers COMT Met/Met Genotype on Placebo vs Healthy Volunteer COMT Val/Val Genotype on Tolcapone vs Healthy Volunteer COMT Val/Met Genotype on Tolcapone vs Healthy Volunteer COMT Met/Met Genotype on Tolcapone; Test type: Other; p = 0.167, ANOVA; Main Effect of Genotype across both Placebo and Tolcapone in left DLPFC

7. Primary Outcome: N-Back Task Activation by Genotype in Patients With Schizophrenia
Description: Activation beta values (N-Back vs. 0-Back) extracted from DLPFC from the contrast maps in Patients with schizophrenia. Lower beta values reflect more efficient processing in the DLPFC when performing working memory tasks.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: 33 patients with schizophrenia
Measure: Mean (Standard Error); unit: beta value
Groups:
- Patients COMT Val/Val Genotype on Placebo: Placebo Days 1-7, Patients COMT Val/Val Genotype
- Patients COMT Val/Met Genotype on Placebo: Placebo Days 1-7, Patients COMT Val/Met Genotype
- Patients COMT Met/Met Genotype on Placebo: Placebo Days 1-7, Patients COMT Met/Met Genotype
- Patients COMT Val/Val Genotype on Tolcapone; Patients COMT Val/Met Genotype on Tolcapone; Patients COMT Met/Met Genotype on Tolcapone: Day 1: Tolcapone 100 mg tid, Days 2-7: Tolcapone 200 mg tid
Arm/Group | Patients COMT Val/Val Genotype on Placebo | Patients COMT Val/Met Genotype on Placebo | Patients COMT Met/Met Genotype on Placebo | Patients COMT Val/Val Genotype on Tolcapone | Patients COMT Val/Met Genotype on Tolcapone | Patients COMT Met/Met Genotype on Tolcapone
Number analyzed (Participants) | 9 | 13 | 11 | 9 | 13 | 11
beta value
  right DLPFC | 0.33 (0.05) | 0.23 (0.03) | 0.24 (0.04) | 0.25 (0.05) | 0.20 (0.03) | 0.22 (0.03)
  left DLPFC | 0.28 (0.04) | 0.24 (0.03) | 0.21 (0.04) | 0.18 (0.05) | 0.26 (0.04) | 0.17 (0.04)
Statistical Analysis 1: Comparison: Patients COMT Val/Val Genotype on Placebo vs Patients COMT Val/Met Genotype on Placebo vs Patients COMT Met/Met Genotype on Placebo vs Patients COMT Val/Val Genotype on Tolcapone vs Patients COMT Val/Met Genotype on Tolcapone vs Patients COMT Met/Met Genotype on Tolcapone; Test type: Other; p = 0.189, ANOVA — Drug by Genotype Effect in left DLPFC
Statistical Analysis 2: Comparison: Patients COMT Val/Val Genotype on Placebo vs Patients COMT Val/Val Genotype on Tolcapone; Test type: Other; p = 0.041, t-test, 1 sided — Drug Effect on Val/Val Genotype in left DLPFC
Statistical Analysis 3: Comparison: Patients COMT Val/Met Genotype on Placebo vs Patients COMT Val/Met Genotype on Tolcapone; Test type: Other; p = 0.718, t-test, 1 sided — Drug Effect on Val/Met Genotype in left DLPFC
Statistical Analysis 4: Comparison: Patients COMT Met/Met Genotype on Placebo vs Patients COMT Met/Met Genotype on Tolcapone; Test type: Other; p = 0.469, t-test, 1 sided — Drug Effect of Met/Met Genotype in left DLPFC

8. Secondary Outcome: Positive and Negative Syndrome Scale
Description: Rating Scales PANSS. The Positive Scale ranges for 7 to 49 with a higher score indicating greater severity of symptoms. The Negative Scale ranges for 7 to 49 with a higher score indicating greater severity of symptoms. The General Scale ranges from 16 to 112, the higher score indicating greater severity of symptoms.
Time Frame: At end of treatment period (at 7th day for first intervention and at 21st day for second intervention)
Population: There were 74 Healthy Volunteers and 33 Patients with Schizophrenia
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Volunteer on Placebo | Healthy Volunteer Tolcapone | Patient on Placebo | Patients on Tolcapone
Number analyzed (Participants) | 74 | 74 | 33 | 33
units on a scale
  Positive Subscale | 7.01 (0.01) | 7.02 (0.03) | 12.15 (0.51) | 12 (0.54)
  Negative Subscale | 7.36 (0.14) | 7.27 (0.13) | 16.51 (1.00) | 15.88 (1.02)
  General Psychopathology | 16.36 (0.10) | 16.33 (0.09) | 27.12 (0.78) | 26.24 (0.84)
Statistical Analysis 1: Comparison: Patient on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.7, t-test, 1 sided — Drug Effect on Positive Syndrome for Patients
Statistical Analysis 2: Comparison: Patient on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.4, t-test, 1 sided — Drug Effect on Negative Syndrome for Patients
Statistical Analysis 3: Comparison: Patient on Placebo vs Patients on Tolcapone; Test type: Other; p = 0.12, t-test, 1 sided — Drug Effect on General Pathology for Patients

ADVERSE EVENTS:
Time Frame: Day 1 to Day 21
Arm/Group | Healthy Volunteers on Placebo | Healthy Volunteers on Tolcapone | Patients on Placebo | Patients on Tolcapone
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/131 | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/131 | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 25/131 | 29/131 | 17/59 | 22/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteers on Placebo (N=131) | Healthy Volunteers on Tolcapone (N=131) | Patients on Placebo (N=59) | Patients on Tolcapone (N=60)
Nausea (Gastrointestinal disorders) | 8 | 16 | 8 | 5 — Nausea was present in two patients in both arms of the protocol.
Sleep Problems (Nervous system disorders) | 8 | 10 | 6 | 17 — Sleep problems was present in three patients in both arms of the protocol.
Appetite Problems (General disorders) | 6 | 8 | 6 | 5 — Appetite problem was present in two patients in both arms of the protocol.
Diarrhea (Gastrointestinal disorders) | 5 | 9 | 4 | 7 — Diarrhea was present in one patient in both arms of the protocol.
Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 6 | 6 | 11 — Stiffness present in four patients in both arms of the protocol.
Halluciantions (Psychiatric disorders) | 0 | 0 | 10 | 9 — Hallucination was present in nine patients in both arms of the protocol. On patient reported hallucinations only on the placebo arm of the protocol.

LIMITATIONS AND CAVEATS:
There was an early termination due to a request from the NIMH leadership to assess if was justifiable to continue when considering costs of this research and needs to assess resources to develop new protocols for the Branch

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes